CLINICAL TRIAL: NCT05720390
Title: Effects of Intragastric Quinine, Alone or Combined With L-leucine, on Postprandial Glycaemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Adelaide (Other)
Responsible Party: Principal Investigator, Christine Feinle-Bisset, Professor, University of Adelaide
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: R20161005-1
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Healthy
Keywords: Intragastric; Quinine; L-leucine; Glycaemic control; Plasma glucose; Glucoregulatory hormones; Gastric emptying; Humans
MeSH Terms: interventions — Quinine; Leucine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In order to blind both investigator and participant, the treatments will be prepared on the morning of each study day, and filled in covered syringes, by a research officer who will have no involvement in data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Quinine only (Active Comparator): In this arm, participants will receive a 10 ml intragastric bolus of 300 mg quinine followed 30 min later by 100 ml intragastric bolus of control for L-leucine.
  Interventions: Other: Quinine; Other: Control
- L-leucine only (Active Comparator): In this arm, participants will receive a 10 ml intragastric bolus of control for quinine followed 30 min later by 100 ml intragastric bolus of 5 g L-leucine.
  Interventions: Other: L-leucine; Other: Control
- Quinine + L-leucine (Active Comparator): In this arm participants will receive a 10 ml intragastric bolus of 300 mg quinine followed 30 min later by 100 ml intragastric bolus of 5 g L-leucine.
  Interventions: Other: Combination of quinine and L-leucine
- Control (Placebo Comparator): In this arm, participants will receive a 10 ml intragastric bolus of control solution followed 30 min later by 100 ml intragastric bolus of control solution.
  Interventions: Other: Control

INTERVENTIONS:
Other: Quinine — Quinine, which is a bitter compound, extracted from the bark of the cinchona tree and has been shown in our previous studies to lower blood glucose in doses of 300-600 mg, will be 'active' in this condition.
  Arms: Quinine only
Other: L-leucine — L-leucine, which is a branched-chain amino acid, and one of the building blocks of protein, therefore is part of our daily diet, will be 'active' in this condition.
  Arms: L-leucine only
Other: Combination of quinine and L-leucine — In this condition, both quinine and L-leucine will be administered as 'active'.
  Arms: Quinine + L-leucine
Other: Control — In the condition, where quinine is 'active', control for L-leucine (5 ml oraplus and 95 ml saline) will be administered. In the condition, where L-leucine will be 'active', control for quinine (10 ml distilled water) will be administered.
  Arms: Control; L-leucine only; Quinine only

SUMMARY:
In this study, participants will receive, in a randomized, double-blind fashion, an intragastric bolus administration of either (i) 300 mg quinine, (ii) 5 g L-leucine, (iii) a combination of (i)+(ii), or (iv) control, before 350 ml (500 kcal) of a mixed-nutrient drink, to evaluate the effects on postprandial blood glucose, gastric emptying, and the hormone responses to the mixed-nutrient drink. Study visits will be separated by 3-7 days and participants will receive one treatment per visit.

On each study visit, the participant will be intubated with a nasogastric feeding tube. At t= - 60 min (08:30 am), a baseline blood sample, visual analogue scale questionnaire (VAS), and breath sample will be collected and quinine or control will be administered through the feeding tube. 30 min later (at t= - 30 min), L-leucine or control will be administered over 2 min after which the feeding tube will be removed immediately. At t = -45, -30, -15, and -1 min further blood samples will be collected and VAS completed. At t = -1 min, participants will consume, within 1 minute, a mixed-nutrient drink, labelled with 100 mg of 1-13C-acetate for measurement of gastric emptying by breath sampling. Blood samples, VAS, and breath samples will be taken at regular intervals between t = 0-180 min.

DETAILED DESCRIPTION:
This trial aims to assess the effects of intragastric administration of quinine, combined with L-leucine, on postprandial blood glucose, gastric emptying, gut and gluco-regulatory hormones, as well as GI symptoms in response to a mixed-nutrient drink.

Each participant will be studied on 4 occasions, separated by 3-7 days. Participants will receive, in randomized, double-blind fashion, an intragastric bolus of (i) 300 mg quinine, (ii) 5 g L-leucine, (iii) combination of (i)+(ii), or (iv) control. Due to the low water solubility, L- leucine will be provided as a suspension using 5 ml of 'the suspending agent' Ora-Plus (manufactured by Perrigo, Minneapolis). Visits will be carried out at the Clinical Research Facility, Adelaide Medical School, University of Adelaide, by staff and students trained in the required clinical research techniques.

Participants will consume a standardized dinner meal (400g McCain's beef lasagne) the night before each study visit by no later than 7 pm. After fasting for 13.5 hours overnight and refraining from alcohol and exercise for 24 hours, participants will arrive at the Clinical Research Facility by 8:30 am. Upon arrival, participants will be intubated with a nasogastric, custom-built soft silicon feeding tube (outer diameter: 4mm; Dentsleeve, Mississauga, Ontario, Canada) that will be inserted through an anaesthetized nostril and placed in the stomach. An intravenous cannula will be placed into a right forearm vein for regular blood sampling. At t = -60 min, a venous baseline blood sample (6 ml) will be collected and the participant will complete a visual analogue scale questionnaire (VAS) to assess GI symptoms (nausea and bloating). Immediately thereafter, the participant will receive a 10- ml intragastric bolus of either 300 mg quinine-hydrochloride (Q-HCl) or water (control), and 30 min later, at t -30 min, an intragastric bolus of L-leucine (100 ml suspension consisting of 5 g L- leucine, 5 ml Ora-Plus and 90 ml 0.9% saline) or control (5 ml Ora-Plus and 95 ml saline) over 1 min after which time the catheter will be removed immediately. At t = -1 min, the participant will consume, within 1 min, a mixed-nutrient drink (Nestle, 500 kcal, 350 ml, 56 g carbohydrates) labelled with 100 mg of 1-13C-acetate for measurement of gastric emptying by breath sampling. Breath samples will be collected in sealed breath bags at baseline (prior to quinine administration) and at regular intervals between t = 0-180 min, for subsequent analysis of 13CO2 concentration in exhaled breath. Blood samples for the measurement of glucose and plasma concentrations of hormones will be taken regularly (12 sampling time points in total), and participant complete VAS questionnaires. At t = 180 min, after final blood and breath samples and VAS measurements, the intravenous cannula will be removed and the participant will be served a light lunch, after which they will be allowed to leave the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Lean weight (BMI 19-25 kg/m2)

Exclusion Criteria:

* Significant gastrointestinal symptoms, disease or surgery;
* Current gallbladder or pancreatic disease;
* Cardiovascular or respiratory diseases;
* Any other illnesses as assessed by the investigator (including chronic illnesses not explicitly listed above);
* Use of prescribed or non-prescribed medications (including vitamins and herbal supplements) which may affect energy metabolism, gastrointestinal function, bodyweight or appetite (eg domperidone and cisapride, anticholinergic drugs (eg atropine), metoclopramide, erythromycin, hyoscine, orlistat, green tea extracts, Astragalus, St Johns Wort etc.);
* Individuals with low ferritin levels (less than 30 ng/mL), or who have donated blood in the 12 weeks prior to taking part in the study;
* Lactose intolerance/other food allergy(ies);
* Vegetarians;
* Restrained eaters (score >12 on the three-factor eating questionnaire);
* Current intake of greater than 2 standard drinks on greater than 5 days per week;
* Current smokers of cigarettes/cigars/marijuana;
* Current intake of any illicit substance;
* High performance athletes;
* Inability to comprehend study protocol;
* Unable to tolerate naso-gastric tube

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline plasma glucose concentration after a mixed-nutrient drink for 3 hours | Blood samples will be taken repeatedly within each study visit (i.e. at baseline (t= 0 minute), after administration of study treatments (t= -45, -30, -15 minutes) and after a mixed-nutrient drink (t= 0, 15, 30, 45, 60, 90, 120 and 180 minutes).
  Plasma glucose concentrations (mmol/L) will be assessed using glucose oxidase method

SECONDARY OUTCOMES:
Gastric emptying of a mixed nutrient drink | Breath samples will be taken repeatedly on each study visit (i.e. t= 0 (baseline), 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 75, 90, 105,120, 135, 150, 165, 180 minutes) to construct a gastric emptying profile on each day.
  Measurement of 13CO2 in breath samples, expressed as percentage of 13CO2 recovery per hour
Plasma concentration of insulin after a mixed-nutrient drink | Blood samples will be taken repeatedly within each study visit (i.e. at baseline (t= 0 minute), after administration of study treatments (t= -45, -30, -15 minutes) and after a mixed-nutrient drink (t= 0, 15, 30, 45, 60, 90, 120 and 180 minutes).
  Plasma insulin concentrations (mU/L) will be assessed using an ELISA immunoassay.
Plasma concentration of glucagon after a mixed-nutrient drink | Blood samples will be taken repeatedly within each study visit (i.e. at baseline (t= 0 minute), after administration of study treatments (t= -45, -30, -15 minutes) and after a mixed-nutrient drink (t= 0, 15, 30, 45, 60, 90, 120 and 180 minutes).
  Plasma glucagon concentrations (pg/mL) will be measured by radioimmunoassay
Gastrointestinal symptoms (nausea and bloating) | Visual Analogue ratings will be collected repeatedly within each study visit (i.e. at baseline (t = 0 minute), after administration of treatments (t= -45, -30, -15 minutes) and after mixed-nutrient drink (t= 0, 15, 30, 45, 60, 90, 120 and 180 minutes).
  Gastrointestinal symptoms will be measured using a 100-mm Visual Analogue Scale (VAS) questionnaire. The minimum value means no feeling at all, and the highest value means feeling very much.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Feinle-Bisset, PhD, Principal Investigator — University of Adelaide, Adelaide, South Australia
Locations (1):
- Clinical Research Facility, Adelaide Health and Medical Sciences Building, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analysed during the current study are not publicly available due to the ethical statement and informed consent that require privacy of data.

REFERENCES:
- [Derived] Sajjad M, Ghorbaninejad P, Bitarafan V, Anjom-Shoae J, Rose BD, Fitzgerald PC, Horowitz M, Feinle-Bisset C. Effects of Combined Intragastric Administration of Quinine with L-Leucine or L-Isoleucine on the Glycemic Response to, and Gastric Emptying of, a Mixed-Nutrient Drink in Healthy Males. J Nutr. 2025 Dec 7:101259. doi: 10.1016/j.tjnut.2025.101259. Online ahead of print. PMID 41365468